CLINICAL TRIAL: NCT02699333
Title: Risk Factors for Microscopic Colitis
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 14-3156
Record Dates: First submitted 2016-02-23; First posted 2016-03-04 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Colitis, Microscopic
MeSH Terms: conditions — Colitis, Microscopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 40 ml of blood centrifuged and separated into plasma, buffy coat and red blood cells. A serum separator tube will be used to collect an additional 10 ml of blood for serum.
  During colonoscopy, four mucosal biopsies will be obtained from normal appearing mucosa in the ascending colon, transverse colon, and descending/sigmoid colon during the withdrawal phase of the exam from each patient (12 research biopsies). To improve orientation 2 biopsies from each segment will be flattened onto filter paper using a forceps and placed together into fixative. The remaining 2 biopsies from each area will be rinsed in sterile PBS to ensure there is no contamination with fecal bacteria prior to freezing in liquid nitrogen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Microscopic colitis cases: Patients found to have microscopic colitis based on colonic biopsies.
- Controls: Patients who meet eligibility requirements but do not have microscopic colitis on biopsy.

SUMMARY:
Microscopic colitis is a common cause of watery diarrhea, particularly in the elderly. Although the incidence is comparable to ulcerative colitis and Crohn's disease, the etiology is unknown. Understanding the etiology of microscopic colitis is an important step in developing logical interventions to decrease the burden from microscopic colitis. This research could provide critical insights into the etiology of this poorly studied condition.

DETAILED DESCRIPTION:
Microscopic colitis (MC) is a chronic condition that is a common cause of watery diarrhea, particularly in the elderly. The etiology is unknown but widely considered to be an abnormal immune reaction to luminal antigens in predisposed hosts. Drugs and autoimmunity have also been implicated. The aims of the study are: 1) To quantitatively classify microscopic colitis using image analysis microscopy to determine whether the degree of lymphocytic infiltration correlates with etiology, symptoms and prognosis. 2) To investigate the etiology of microscopic colitis by examining medical and lifestyle risk factors including medications, autoimmunity, diet, and smoking 3) To evaluate the association between the adherent microbial flora and MC to assess whether bacterial dysbiosis is linked to presence of MC. As an exploratory aim we will evaluate whether CYP2C19 polymorphisms are more common in purportedly drug-induced disease since the diverse drugs that have been associated with MC are all substrates for this gene.

To conduct the study the investigators will obtain detailed dietary, medical and lifestyle information on study subjects who undergo complete colonoscopy for diarrhea. The investigators will obtain colon biopsies from the right, transverse and left colon to evaluate adherent bacterial organisms. The investigators will draw blood to evaluate CYP2C19 polymorphisms and for future genetic studies. The prospective design corrects important limitations of prior research on MC. Successful completion of the study aims will improve the understanding of risk factors, set the stage for more scientifically grounded future research, and potentially suggest new interventions for a disease that is currently poorly understood.

ELIGIBILITY:
Inclusion Criteria:

Colonoscopy for diarrhea

Exclusion Criteria:

1. Fewer than 4 loose bowel movements per day.
2. Failure to visualize the entire colon to the cecum or preparation less than good or excellent.
3. Age under 35 years. There will be no upper age limit.
4. Inability to understand and cooperate with the interview.
5. Indication for colonoscopy other than diarrhea.
6. Prior history of inflammatory bowel disease (Crohn's disease or ulcerative colitis).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo colonoscopy for diarrhea at the University of North Carolina
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Microscopic Colitis | Day 1
  Microscopic colitis defined by increased lymphocytes or collagen

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Sandler, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided